CLINICAL TRIAL: NCT04049149
Title: Precision Medicine to Redefine Insulin Secretion and Monogenic Diabetes (PRISM) in Chinese Patients With Young Onset Diabetes
Brief Title: Precision Medicine in Chinese Patients With Young Onset Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CRE-2019.080
Record Dates: First submitted 2019-07-22; First posted 2019-08-07 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Type 2 Diabetes
Keywords: Young-onset type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JADE-PRISM group (Other): Only applicable in part 3 which is a randomized controlled trial. Part 1 and part 2 are the prospective cohort studies.
  Interventions: Other: Biogenetic explanation and endocrinologist intensive managment
- JADE group (Other): Only applicable in part 3 which is a randomized controlled trial. Part 1 and part 2 are the prospective cohort studies.
  Interventions: Other: Usual care management

INTERVENTIONS:
Other: Biogenetic explanation and endocrinologist intensive managment — * JADE report and JADE APP
  * Biogenetic explanation
  * First-year intensive management by endocrinologists
  * Follow up by their usual care doctors for continue treatment regimen maintenance.
  * Yearly DM nurses follow up for blood taking and questionnaires
  Arms: JADE-PRISM group
Other: Usual care management — * JADE report and JADE APP
  * Attend their usual care clinic for ongoing treatment
  * Yearly DM nurses follow up for blood taking and questionnaires
  Arms: JADE group

SUMMARY:
Patients with young onset diabetes (YOD) are one of the most challenging groups of patients due to their long disease duration, complex causes, delayed interventions, psychosocial stress, poor adherence and frequent default. The investigator's previous studies indicate that provision of biogenetic information improved satisfaction, reduced ambiguity and improved self-efficacy in patients with T2D. Provision of personalized information using the web-based Joint Asia Diabetes Evaluation (JADE) Technology with risk stratification and decision support empowers better self care and medical intervention with improved control of risk factors. To further improve the precision of diagnosis for individualizing care, the use of CP, GADA, genetic risk scores (GRS) or rare genetic variants of maturity onset of diabetes (MODY) can help doctors select the most appropriate therapy in a timely manner. While patients with low CP, GADA and high GRS will benefit from early insulin therapy, some MODY variants are associated with good response to insulin-releasing oral drugs (e.g. sulphonylurea) which may spare the use of insulin with reduced patient distress and over-insulinization. By contrast, patients with high CP often due to obesity-associated insulin resistance should undergo intensive lifestyle modification and use of drugs with weight-reducing or neutral effects to avoid weight gain due to excessive dose of insulin.

DETAILED DESCRIPTION:
Patients with young onset diabetes (YOD) are one of the most challenging groups of patients due to their long disease duration, complex causes, delayed interventions, psychosocial stress, poor adherence and frequent default. The investigator's previous studies indicate that provision of biogenetic information improved satisfaction, reduced ambiguity and improved self-efficacy in patients with T2D. Provision of personalized information using the web-based Joint Asia Diabetes Evaluation (JADE) Technology with risk stratification and decision support empowers better self care and medical intervention with improved control of risk factors. To further improve the precision of diagnosis for individualizing care, the use of CP, GADA, genetic risk scores (GRS) or rare genetic variants of maturity onset of diabetes (MODY) can help doctors select the most appropriate therapy in a timely manner. While patients with low CP, GADA and high GRS will benefit from early insulin therapy, some MODY variants are associated with good response to insulin-releasing oral drugs (e.g. sulphonylurea) which may spare the use of insulin with reduced patient distress and over-insulinization. By contrast, patients with high CP often due to obesity-associated insulin resistance should undergo intensive lifestyle modification and use of drugs with weight-reducing or neutral effects to avoid weight gain due to excessive dose of insulin.

PART 1:

Objective: To characterize Chinese patients diabetes classified by fasting CP and GADA positivity and their prognostic significance.

Methods: Fasting CP levels and GADA in stored biosamples of 4000 patients in the Hong Kong Diabetes Register (HKDR) followed up since 1995.

PART 2:

Objective: To uncover genetic variants/sequences associated with familial YOD. Methods: Whole genome sequencing (WGS) in stored DNA of 100-120 sibpairs of YOD after 13 years of follow-up for imputation with exome data of case-control cohort of YOD and genome wide association studies (GWAS) data of 200 YOD families and 6000 T2D patients.

PART 3:

Objectives: To examine the impacts of precision medicine augmented by information technology and biogenetic markers (JADEPRISM) on attainment of cardiometabolic targets at 1 year and clinical outcomes at 3 year (n=440), compared with JADE-augmented care (n=440) in YOD.

Deliverables A catalogue of biogenetic markers to guide precision medicine augmented by the JADE-Technology to optimize clinical outcomes in YOD.

ELIGIBILITY:
Inclusion Criteria:

Part 1: Prospective cohort of Chinese with type 2 diabetes

Between 1995 and December 2004, 10,129 patients were assessed using structured protocol to esetablish the HKDR and of them, we have measured GADA and CP in 1400 patients with YOD. In this study, we shall measure CP and GADA in 4000 subjects from the HKDR with available GWAS data irrespective of their age of diagnosis. These samples were linked to our various databases by a unique identification code which will enable us to track the clinical outcomes including development of complications.

Part 2: Family-based cohort of first-degree relatives of diabetic probands

We shall utilize the resource of the HKDFS and control subjects to discover novel genetic variants of YOD. Subjects will be selected based on their status with or without diabetes. In 2012-2013, we ascertained the glycemic status of 365 siblings in the HKDFS and 452 participants of the community-based LKS cohort (aged 18-55 years) without diabetes at baseline (1998-2002).

In this cohort, 167 participants (53.7%) with a family history of YOD, 68 participants (30.1%) with a family history of late onset diabetes and 40 (14.4%) participants without family history of diabetes developed diabetes. Amongst the 313 siblings with family history of YOD, 167 had diabetes at baseline or developed diabetes during follow up and 146 did not develop diabetes after 13 years giving 100-120 sibpairs for linkage analysis. These sequence data will be imputed with 500 YOD patients and 500 control subjects with exome data as well as 6000 patients in the HKDR with GWAS data for analysis for validation purpose.

Part 3: RCT (PRISM)

* Non-type 1 diabetes (T1D)
* Chinese ethnicity
* Age between 18-50 years inclusive
* Age at diabetes diagnosis 40 years
* Able to understand study requirements and voluntarily agree to participate by providing written informed consent

Exclusion Criteria:

Part 1/2:

Subjects in the HKDR, HKFDS and LKS cohorts without or insuffiicent amount of biosamples for assays or sequencing.

Part 3:

* T1D, defined by presentation with diabetic ketoacidosis or insulin requirement within 6 months of diagnosis.
* Reduced life expectancy due to terminal illness or otherwise deemed not appropriate per discretion of the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 884 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of C-Peptide (CP) and Glutamic Acid Decarboxylase Antibody (GADA) in Chinese adult patients with T2D (Part 1 of study) | through study completion, an average of 4 years
  Between 1995 to 2004, all patients in the HKDR had structured assessment with storage of blood samples (collected at registration) for future research purpose. We shall measure CP and GADA in 4000-5000 patients.
The correlation of C-Peptide (CP) and Glutamic Acid Decarboxylase Antibody (GADA) on clinical outcomes (Part 1 of study) | through study completion, an average of 4 years
  Between 1995 to 2004, all patients in the HKDR had structured assessment with storage of blood samples (collected at registration) for future research purpose.
Incidence of young-onset type 2 diabetes and its genetic susceptibility (Part 2 of study) | through study completion, an average of 4 years
  Between 1998 to 2013, subjects from the HKFDS and the community-based LKS cohort had storage of blood samples at registration.
Incidence of any diabetes-related micro/macrovascular endpoints (Part 3 of study) | through study completion, an average of 4 year
  Incident including cardiovascular disease (coronary heart disease, congestive heart failure, stroke, peripheral artery disease), chronic kidney disease, all-cause death and/or incident/progression/remission of albuminuria, estimated glomerular filtration rate, retinopathy, visual acuity and sensory neuropathy

SECONDARY OUTCOMES:
The levels of CP and GADA and the number of genetic variants for disease prognositication and classification to guide precision medicine in YOD (Part 1 and 2 of study) | through study completion, an average of 4 years
The number of genetic variants for disease prognositication and classification to guide precision medicine in YOD (Part 1 and 2 of study) | through study completion, an average of 4 years
The number of novel targets and pathways for discovery of drug targets with companian diagnostics (Part 1 and 2 of study) | through study completion, an average of 4 years
The number of patients attaining ≥3 cardiometabolic risk factors (Part 3 of study) | through study completion, an average of 4 years
  Defined as A1c<6,2%, blood pressure<120/80 mmHg, LDL-C<1.8 mmol/L , triglyceride<1.2 mmol/L, waist circumference<80 cm in women <85 cm in men which has been shown to reduce cardiovascular-renal endpoint in the JDOIT- 3 Study compared to conventional targets (A1c<7%, BP<130/80, LDL-C<1.8 mmol/L, triglyceride <1.7 mmol/L)
Incidence of severe hypoglycaemia (Part 3 of study) | through study completion, an average of 4 year
  Defined as hospitalization due to hypoglycaemia
Rate of changes in glycaemic control (Part 3 of study) | through study completion, an average of 4 year
  changes in HbA1c
On-treatment changes in blood pressure (Part 3 of study) | through study completion, an average of 4 year
  measure both systolic and diastolic blood pressure in mmHg
On-treatment changes in lipid profiles (Part 3 of study) | through study completion, an average of 4 year
  measure the changes in Total cholesterol, Triglyceride, High-density lipo-protein cholesterol, Low-density lipo-protein cholesterol
On-treatment changes in Body Mass Index (Part 3 of study) | through study completion, an average of 4 year
  Measure by BW in kg
On-treatment changes in CP (Part 3 of study) | through study completion, an average of 4 year
  Measure by changes in C-peptide
Rate of changes in use of medications (Part 3 of study) | through study completion, an average of 4 year
Changes in patient's Quality of life (Part 3 of study) | through study completion, an average of 4 year
  Measure by questionnaire: EQ-5D For Quality of life (Total 5 questions with total score 1-15, highest score indicates the worst outcome)
Changes in patient's reported outcomes : Depression (Part 3 of study) | through study completion, an average of 4 year
  Measure by questionnaire: PHQ-9 For Depression (Total 9 questions with total score 0-27, highest score indicates the worst outcome)
Changes in patient's compliance (Part 3 of study) | through study completion, an average of 4 year
  Measure by questionnaire: CQ-4 For Compliance (Total 4 questions with total score 0-4, highest score indicates the worst outcome)
Changes in patient's diabetes empowerment (Part 3 of study) | through study completion, an average of 4 year
  Measure by Diabetes Empowerment Scale (DES-20 for efficacy) (Total 20 questions with total score 0-80, highest score indicates better outcome)
Changes in patient's diabetes self care activities (Part 3 of study) | through study completion, an average of 4 year
  Measure by questionnaire: Summary of diabetes self care activities (SDSCA-15 For self care) (Total 15 questions with total score 0-105, highest score indicates better outcome)
Changes in patient's perceived personal control (Part 3 of study) | through study completion, an average of 4 year
  Measure by Perceived personal control (PPC) questionnaire (Total 9 questions with total score 0-18, highest score indicates better outcome)
Changes in patient's genetic counseling satisfaction (Part 3 of study) | through study completion, an average of 4 year
  Measure by Genetic counseling satisfaction scale (GCSS) (Total 6 questions with total score 1-30, highest score indicates better outcome)
Changes in patient's diabetes related distress (Part 3 of study) | through study completion, an average of 4 year
  Measures by questionnaire: Diabetes Distress Scale (DDS; total score from 17-102), comprising 3 subscales namely emotional, physician, regimen / social support. A lower score indicates better outcome
Changes in patient's Depression Anxiety Stress (Part 3 of study) | through study completion, an average of 4 year
  Measure by Depression Anxiety Stress Scale (DASS-21) (Total 21 questions with total score 0-63, lowest score indicates better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Derived] O CK, Fan YN, Fan B, Lim C, Lau ESH, Tsoi STF, Wan R, Lai WY, Poon EW, Ho J, Ho CCY, Fung C, Lee EK, Wong SY, Wang M, Ozaki R, Cheung E, Ma RCW, Chow E, Kong APS, Luk A, Chan JCN. Precision Medicine to Redefine Insulin Secretion and Monogenic Diabetes-Randomized Controlled Trial (PRISM-RCT) in Chinese patients with young-onset diabetes: design, methods and baseline characteristics. BMJ Open Diabetes Res Care. 2024 Jun 19;12(3):e004120. doi: 10.1136/bmjdrc-2024-004120. PMID 38901858